CLINICAL TRIAL: NCT01453881
Title: Randomized Clinical Trials to Compare Asthma Control Efficacy of the Fine-particle Combination Formoterol/Beclomethasone by pMDI Administered With and Without Spacer.
Brief Title: Fine Particle pMDI Formoterol/Beclomethasone in Asthmatics With and Without Spacer: Comparative Efficacy Evaluation
Acronym: EFFECT-EV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Universidade Federal do vale do São Francisco (Other)
Responsible Party: Principal Investigator, Jose Angelo Rizzo, PhD, MD, Medicine Professor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTC 034/11
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Asthma
Keywords: Asthma; pMDI; Beclomethasone; Formoterol; Efficacy
MeSH Terms: conditions — Asthma | interventions — Metered Dose Inhalers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spacer (Experimental): Beclomethasone/Formoterol 100/6mcg/puff pMDI 2 puffs two times/day with the aid of a Valved Holding Chamber - VORTEX
  Interventions: Device: Spacer
- Comparator (Active Comparator): Beclomethasone/Formoterol pMDI 100/6mcg/puff pMDI 2 puffs two times/day without the aid of a Valved Holding Chamber - VORTEX
  Interventions: Device: Comparator

INTERVENTIONS:
Device: Spacer — Beclomethasone/Formoterol 100/6mcg pMDI 2 puffs two times/day with the aid of a Valved Holding Chamber - VORTEX
  Other Names: BECLOMETHASONE EXTRA-FINE; FORMOTEROL; FOSTAIR; INNOVAIR; VORTEX
  Arms: Spacer
Device: Comparator — Beclomethasone/Formoterol 100/6mcg pMDI 2 puffs two times/day without the aid of a Valved Holding Chamber - VORTEX
  Arms: Comparator

SUMMARY:
Adequate pharmacological treatment controls symptoms in most asthmatics. Pressurized metered dose inhalers (pMDI)are the most used drug delivery devices. Valved holding chambers of different types and sizes have also been developed for use in combination with pMDI. The therapeutic efficacy of treatment depends on the amount of inhaled particles. The chambers can optimize lung deposition as it obviates lung-hand coordination and retain larger particles. The aim of this study is to compare the efficacy of the fine particle combination pMDI Beclomethasone/Formoterol in asthma control,with or without the aid of a spacer in patients without adequate asthma control on medium to high-dose inhaled steroids associated with long acting beta adrenergic drugs. The hypothesis is that there is no clinical efficacy difference between the two forms of drug administration.

DETAILED DESCRIPTION:
This is a randomized, parallel controlled study with blind outcome evaluation to compare the efficacy of the fine particle combination Beclomethasone/Formoterol administered with or without valved holding chamber (Vortex, Pari Innovative Manufacturers, VA - USA.

Eligible asthma patients will begin a 2-weeks run-in period to optimize their control medication use and to learn the correct relief pMDI use without holding chamber. After the run-in, patients with non-controled asthma symptoms (ACT score 19 or under)in spite the use of medium to high dose inhaled steroids and LABA association and able to use correctly the pMDI will be randomized (block-randomization) to receive the test medication combination to be used with or without the spacer device (VORTEX). Patients will be evaluated after 30 and 60 days. At days 15 (+,- 2) and 45 (+,- 2) they will have an incentive phone call.

ACT score (translated and validated to portuguese - Brazil), FEV1 (Kit-Micro spirometer, Cosmed, Italy), pMDI use and clinical evaluation will be obtained at initial visit (visit 0), randomization visit (visit 1)and at 30 and 60 days (visits 2 and 3). Extra-medication allowed at run-in period will be inhaled beta-2 bronchodilators for relief an at treatment period inhaled beta-2 agonists for relief and systemic steroids for exacerbations, with antibiotics as needed.

Endpoint evaluations will be proceeded by a treatment blinded investigator.In order to keep the concealment, the evaluations will be held in a different room and the patients instructed not to comment on treatment.

Subjects will be excluded at the treatment period in case of severe asthma exacerbation (hospital or ICU recovery or systemic steroid used for more than 5 days). They will be excluded also in case of concomitant ailments at discretion of the attending physician. These patients will be excluded from the per-protocol evaluation but will be described.

Sample size was calculated taking into account a relevant ACT score difference of 3 points and a SD of 4.4 (SCHATZ M et all. Asthma Control Test: reliability, validity, and responsiveness in patients not previously followed by asthma specialists. J Allergy Clin Immunol 2006;117:549-56). In order to be able to detect this difference with α and β errors of 5% and 20% respectively, the investigators calculated 32 patients per group.

Statistical analysis will be carried according to data distribution by a professional statistician.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, age 18 to 65 years, both sexes;
2. Clinical diagnosis of moderate to severe persistent asthma;
3. Nonsmoker;
4. Agree to participate and sign the Informed Consent;
5. ACT Score <= 19
6. FEV1 <= 80% of predicted;
7. History of response to FEV1 greater than 10%;
8. Patients who are already using Inhaled steroids at medium to high doses (Beclomethasone, budesonide, fluticasone) with longa-acting beta2 agonists (formoterol or salmeterol)
9. Proper use of metered-dose inhaler (after orientation)

Exclusion Criteria:

1. Patient diagnosed with Chronic Obstructive Pulmonary Disease (COPD);
2. Current smokers or have stopped for less than 10 years;
3. Patients with a history of recent near-fatal asthma (less than 12 months);
4. Patients with a history of recent asthma hospitalization (last 6 months);
5. Patients with airway infection symptoms for less than 4 weeks;
6. Participation in any experimental study up to 1 (one) year from selection visit;
7. Hospitalization for any reason up to 8 weeks before selection visit;
8. History of liver, cardiac, renal, pulmonary or gastrointestinal diseases, epileptic, psychiatric or hematologic disorders, uncontrolled hypertension, rheumatology/orthopedic disorders that interferes with pMDI use;
9. Patients unable to properly use the pMDI during the selection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in Asthma Control Test Score | 8 weeks
  The primary endpoint is the difference in the change of ACT score between groups 8 weeks after randomization compared to pre-randomization.

SECONDARY OUTCOMES:
Changes in Forced Expiratory Volume in the first second (FEV1) | 4 and 8 weeks
  The secondary endpoint is the difference in the change on FEV1 between groups at 4 and 8 weeks after randomization compared to pre-randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Rizzo, PhD, MD, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Hospital das Clínicas - Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil